CLINICAL TRIAL: NCT03040700
Title: "Long-term Follow-up of Patients With Multivessel Coronary Artery Disease Undergoing CABG - Comparison Between Functional, Anatomical, or Medical Only-Based Evaluation to Prevent Cardiovascular Events - The FAMOUS Trial"
Brief Title: Follow-up of Patients With Multivessel Coronary Artery Disease After CABG
Acronym: FAMOUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Luis Henrique W Gowdak, MD, PhD, Clinical Scientist, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 405153/2012-0
Record Dates: First submitted 2017-01-06; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Coronary (Artery); Disease
Keywords: coronary artery disease; surgery; angina; myocardial ischemia; non-invasive testing
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clinical (No Intervention): Regular medical visits every 6 months.
- Myocardial Perfusion Scan (Experimental): Myocardial perfusion stress test using cardiac scintigraphy (Sestamibi) at rest and during pharmacological stress (dipyridamole)
  Interventions: Other: Myocardial Perfusion Scan
- Coronary CTA (Experimental): Coronary computed tomography angiography
  Interventions: Other: Coronary CTA

INTERVENTIONS:
Other: Myocardial Perfusion Scan — Myocardial perfusion scan will be performed at rest and during pharmacological stress with dipyridamole (99mTc-Sestamibi)
  Arms: Myocardial Perfusion Scan
Other: Coronary CTA — Coronary CTA will be performed using a 320-detector scanner, 0.5 mm slice thickness, with gantry rotation of 350ms. Prior to each scan, the patient's blood pressure and heart rate will be assessed, and if the heart rate is above 70bpm, beta-blockers will be given orally. Following oral beta blocker administration, if the heart rate is still greater than 64bpm, intravenous metoprolol will be administered. A total of 70-100 mL of iodinated contrast will be administered via an automated injector at a rate of 5mL/s. All coronary CTA images will be transferred to a workstation (Vitrea FX-Vital Image) and analyzed by two experienced cardiac imagers who are blinded to all other data using a standard 18-segment coronary tree model.
  Arms: Coronary CTA

SUMMARY:
The FAMOUS Trial is a single-center, prospective, randomized study aimed to compare three different strategies (clinical, anatomical, or functional) in preventing MACE after CABG. A total of 600 patients will be included and followed for 5 years. Patients will be randomly allocated (1:1:1) in one of the three follow-up strategies. Patients in the clinical arm will be followed by regular medical visits only every 6 months; patients in the functional arm will undergo a myocardial perfusion scan, and those in the anatomical arm will be subjected to a coronary CT. Non-invasive tests will be performed per protocol and regardless symptoms every 2 years after the first year post-surgery. The primary outcome will be the incidence of death, acute myocardial infarction or myocardial revascularization.

DETAILED DESCRIPTION:
Background: Coronary artery disease (CAD) is a highly prevalent clinical condition, usually associated with impairment in quality of life, and with a high risk for cardiovascular events including myocardial infarction and cardiovascular death. Because of the anatomical and/or functional extension of the disease, combined with high-risk clinical features (left ventricular dysfunction, diabetes, or chronic kidney disease to name a few), many patients must undergo a coronary artery bypass grafting (CABG) surgery. In the USA, 400,000 CABG surgeries are performed annually.

Although the benefits of CABG for those high-risk patients have been well established in the long-term, the best follow-up strategy after surgery is still controversial. Current guidelines generally recommend that the follow-up of patients after CABG should be based on the same strategies proposed for patients with stable angina. The investigators hypothesized that the early identification of myocardial ischemia or progression of coronary atherosclerosis, even in asymptomatic patients, may be superior to clinical follow-up alone for the prevention of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Documented obstructive coronary artery disease
* Isolated, recent CABG (< 30 days from inclusion)

Exclusion Criteria:

* Concomitant, severe heart disease from other etiologies including valvular heart disease, advanced dilated cardiomyopathy, etc
* Glomerular filtration rate < 30mL/min/1.73m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Composite fatal/non-fatal MACE | 5 years post-CABG
  All-cause death, non-fatal MI, or myocardial revascularization

SECONDARY OUTCOMES:
Cardiovascular death | 1, 3, and 5 years post-CABG
  Death related to cardiovascular events including sudden death, and death due to acute coronary syndromes (unstable angina, myocardial infarction), heart failure, myocardial revascularization procedures
Cardiovascular hospitalizations | 1, 3, and 5 years post-CABG
  Hospital admissions due to cardiovascular events

OTHER OUTCOMES:
Angina functional class | 1, 3, and 5 years post-CABG
  Canadian Cardiovascular Society classification of angina
Left ventricular function | 1, 3, and 5 years post-CABG
  LV ejection fraction assessed by echocardiography
Decline in renal function | 1, 3, and 5 years post-CABG
  Assessment of the GFR by the MDRD Equation
Incidence of cancer | 1, 3, and 5 years post-CABG
  Incidence of any, new diagnosed cancer

CONTACTS AND LOCATIONS:
Overall Officials: Luis Henrique W Gowdak, MD, PhD, Principal Investigator — Heart Institute
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No